CLINICAL TRIAL: NCT00740389
Title: A Phase I, Open-label Trial to Investigate the Pharmacokinetic Interaction Between TMC125 and Two Antifungal Agents (Fluconazole and Voriconazole), All at Steady-state in Healthy Subjects.
Brief Title: TMC125-TiDP2-C187: A Phase I, Open-label Trial to Investigate the Pharmacokinetic Interaction Between TMC125 and Two Antifungal Agents (Fluconazole and Voriconazole), All at Steady-state in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR014992
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-04

CONDITIONS: HIV; AIDS; Fungal Infection
Keywords: TMC125-C187; TMC125-TiDP2-C187; HIV; AIDS; Fungal Infection; Pharmacokinetics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Mycoses | interventions — etravirine

INTERVENTIONS:
Drug: TMC125

SUMMARY:
This is a Phase I, open-label, 3-period crossover trial to investigate the pharmacokinetic interaction (process by which a drug is absorbed, distributed, metabolised and eliminated by the body) between TMC125 and fluconazole, and between TMC125 and voriconazole.

DETAILED DESCRIPTION:
In this Phase I, open-label, 3-period crossover trial the potential pharmacokinetic interaction between TMC125 and fluconazole and between TMC125 and voriconazole will be investigated. Fluconazole and voriconazole are triazole antifungal agents.

Fluconazole and voriconazole are inhibitors of CYP isoenzymes 2C19, 2C9 and CYP3A4. Fluconazole is metabolized by the liver to a small extent. Approximately 80% of the administered fluconazole dose appears in the urine in unchanged form. Voriconazole is metabolized by CYP2C19, 2C9 and 3A4. TMC125 is also metabolized by CYP3A, 2C9 and 2C19. Because of the effect of fluconazole and voriconazole on the metabolic pathways relevant for TMC125 metabolism, concomitant administration of TMC125 and fluconazole or voriconazole might increase TMC125 pharmacokinetics. Because of the effect of TMC125 on the metabolic pathways relevant for voriconazole metabolism, concomitant administration of TMC125 and voriconazole might also modify voriconazole pharmacokinetics. Since the elimination of fluconazole is mainly via the kidneys, an effect of TMC125 on fluconazole pharmacokinetics is not expected. The current trial aims to assess the 2-way pharmacokinetic interaction between TMC125 and fluconazole, and between TMC125 and voriconazole, to provide dosing recommendations for combined use in the treatment of HIV infected patients.In this trial the pharmacokinetic interaction between TMC125 and fluconazole, and between TMC125 and voriconazole, all at steady-state will be investigated in 18 healthy subjects. During the first two sessions, each subject will receive 2 treatments (Treatments A and B) in a randomized way. In Treatment A, 200 mg TMC125 twice a day. will be administered from Day 1 to Day 7 with an additional morning dose on Day 8. In Treatment B, 200 mg fluconazole once a day in the morning will be administered from Day 1 to Day 16, co-administered with 200 mg TMC125 twice a day from Day 9 to Day 16.

These sessions are followed by a third session, Treatment C, in which 400 mg voriconazole twice a day will be administered on Day 1 and 200 mg voriconazole twice a day will be administered from Day 2 to Day 15, with an additional morning dose on Day 16. From Day 9 to Day 15, 200 mg TMC125 twice a day will be co-administered, with an additional morning dose on Day 16. All TMC125 and fluconazole intakes will be under fed conditions, within 10 minutes after a meal. Voriconazole will be administered 1.5 hour before a meal. Between subsequent treatment sessions, there will be a washout period of at least 2 weeks. Full pharmacokinetic profiles will be determined for one dosing interval (12 hours) for TMC125 on Day 8 of Treatment A and on Day 16 of Treatments B and C. For fluconazole, full pharmacokinetic profiles will be determined for one dosing interval (24 hours) on Days 8 and 16 of Treatment B. For voriconazole, full pharmacokinetic profiles will be determined for one dosing interval (12 hours) on Days 8 and 16 of Treatment C. Safety and tolerability will be monitored continuously throughout the trial. Treatment A: 200 mg TMC125 twice daily, orally from Day 1 to 7 and a morning dose on Day 8. Treatment B: 200 mg fluconazole once daily, orally from Day 1 to 16, co-administered with 200 mg TMC125 twice daily from Day 9 to 16. Treatment C: 400 mg voriconazole twice daily, orally on Day 1 and 200 mg voriconazole twice daily will be administered from Day 2 to 15, with a morning dose on Day 16. From Day 9 to 15, 200 mg TMC125 twice daily will be co-administered, with a morning dose on Day 16.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to screening
* Body Mass Index (BMI) of 18.0 to 30.0 kg/m2, extremes included. BMI is calculated as the weight (in kg) divided by the square of height (in m)
* Informed Consent Forms signed voluntarily before first trial-related activity
* Able to comply with protocol requirements
* Healthy on the basis of medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination (including skin examination), medical and surgical history, electrocardiogram (ECG), vital signs and the results of blood biochemistry, hematology and a urinalysis carried out at Screening.

Exclusion Criteria:

* A positive HIV-1 or HIV-2 test at study screening
* Female, except if postmenopausal since more than two years, or post-hysterectomy or surgically sterilized (without reversal operation)
* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use which in the investigator's opinion would compromise subject's safety and/or compliance with study procedures
* Hepatitis A infection, hepatitis B infection, or hepatitis C infection at study screening
* A positive urine drug test at study screening or on Day -1 of each session. Urine will be tested for the presence of amphetamines, benzodiazepines, cocaine, cannabinoids and opioids
* Currently active or underlying gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory or infectious disease
* Currently significant diarrhea, gastric stasis or constipation that in the investigator's opinion could influence drug absorption or bioavailability
* Any history of significant skin disease. Previously demonstrated clinically significant allergy or hypersensitivity to fluconazole, voriconazole and/or any of the excipients of the investigational medication administered in this trial
* Clinical evidence or history of long QT syndrome and history of additional risk factors for Torsade de Pointes, such as cardiomyopathy, heart failure, hypokalemia, family history of known Long QT Syndrome, or sudden unexplained death at a young age (= 40 years) in a firstdegree relative (i.e., biological parent, sibling, or offspring)
* Clinically relevant heart rhythm disturbances known or suggested by history, or on 12-lead ECG at screening or on Day 1 (predose) of the first treatment period
* Electrolyte abnormalities (hypokalemia, hypocalcemia, hypomagnesemia), grade 2 or greater, within 21 days prior to intake of the investigational medication
* History of galactose intolerance, lactase deficiency or glucose-galactose malabsorption
* Use of concomitant medication, including over-the-counter products and dietary supplements
* Systemic over-the-counter medication must have been discontinued at least 7 days prior to the first dose of study medication
* prescribed medication and all products containing Hypericum perforatum (e.g. St. John's wort) must have been discontinued at least 14 days before the first dose of study medication, except for paracetamol
* Participation in an investigational drug trial within 60 days prior to the first intake of trial medication
* Donation of blood or plasma within the 60 days preceding the first drug intake
* Having participated in more than 1 trial with TMC125 (etravirine), TMC120 (dapirivine) and/or TMC278 (rilpivirine, formerly known as R278474) or having developed rash, erythema or urticaria while participating in a trial with the aforementioned compounds
* Subjects with the laboratory abnormalities at screening as defined by the Division of AIDS and in accordance with the normal ranges of clinical laboratory.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of TMC125, voriconazole and fluconazole

SECONDARY OUTCOMES:
short-term safety and tolerability of the coadministration of voriconazole or fluconazole and TMC125

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- [Derived] Kakuda TN, Van Solingen-Ristea R, Aharchi F, Smedt GD, Witek J, Nijs S, Vyncke V, Hoetelmans RM. Pharmacokinetics and short-term safety of etravirine in combination with fluconazole or voriconazole in HIV-negative volunteers. J Clin Pharmacol. 2013 Jan;53(1):41-50. doi: 10.1177/0091270011433329. Epub 2013 Jan 24. PMID 23400742
- See also: Clinical Study Report Synopsis of TMC125-TiDP2-C187: A Phase I, open-label trial to investigate the pharmacokinetic interaction between TMC125 and two antifungal agents (fluconazole and voriconazole), all at steady-state in healthy volunteers. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1009&filename=CR014992_CSR.pdf